CLINICAL TRIAL: NCT03745560
Title: Simultaneous Translabyrinthine Surgery of Vestibular Schwannoma and Cochlear Implantation with Intraoperative EBERA and Correlation to Hearing Results - a Pilot Study
Brief Title: Intraoperative EABR for Decision Making
Status: Recruiting | Type: Observational
Sponsor: Christoph Arnoldner (Other)
Responsible Party: Sponsor-Investigator, Christoph Arnoldner, Assoc. Prof PD. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1111/2017
Record Dates: First submitted 2018-11-03; First posted 2018-11-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Vestibular Schwannoma; Hearing Loss
Keywords: Cochlear implant
MeSH Terms: conditions — Neuroma, Acoustic; Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study patients undergoing simultaneous translabyrinthine vestibular schwannoma resection and cochlear implantation are included. The goal of the study is to correlate the eABR results with postoperative hearing results.

DETAILED DESCRIPTION:
Patients undergoing translabyrinthine vestibular schwannoma resection are included in the study. Preoperatively an eABR is carried out, as well as before and after tumor resection.

Postoperatively patients are fitted with a cochlear implant as routinely carried out. The postoperative hearing results with cochlear implant are correlated to the eABR results. The study is an observational study since eABR measurements are not part of the study. A correlation between eABR results categorized in three groups (good response, weak response, no response) with monosyllable understanding with cochlear implant (measured with Freiburger monosyllables test).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 99 years undergoing translabyrinthine vestibular schwannoma resection
* Patients wanted hearing rehabilitation with a cochlear implant

Exclusion Criteria:

* patients who do not want to be part of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing translabyrinthine vestibular schwannoma resection and cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Correlation of eABR results to postoperative hearing results | 2 years
  eABR is correlated with postoperative hearing results eABR will be divided in three categories - good response, weak response, no response.
  Hearing results will be measured with speech understanding in Freiburg monosyllables word test which is measured in % of monosyllables understanding at 65 and 80dB

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Arnoldner, MD, Principal Investigator — MUW, Allgemeines Krankenhaus
Locations (1):
- AKH, MUW, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gadenstaetter AJ, Auinger AB, Gerlitz M, Riss D, Yildiz E, Roessler K, Matula C, Dahm V, Arnoldner C. Long-Term Follow-Up After Translabyrinthine IAC Tumor Removal With Simultaneous Cochlear Implantation. Otol Neurotol. 2025 Dec 1;46(10):1310-1315. doi: 10.1097/MAO.0000000000004313. Epub 2025 Nov 12. PMID 39284021